CLINICAL TRIAL: NCT05378620
Title: Project Dulce for Filipino-Americans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22-7886; KL2TR002552 (NIH)
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Type 2
Keywords: Diabetes; Self-Management; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project Dulce + Dulce Digital (Other): Patients will participate in a peer-led group diabetes self-management education and support program and receive ongoing support via text messages designed to improve knowledge, health beliefs, self-management behaviors and clinical outcomes.
  Interventions: Behavioral: Project Dulce + Dulce Digital

INTERVENTIONS:
Behavioral: Project Dulce + Dulce Digital — Project Dulce will consist of a group diabetes self-management program consisting of a 5-week curriculum delivered by a peer educator in Tagalog. The curriculum provides new knowledge as well as skills and tools needed to adapt to a life with diabetes and change behaviors. The curriculum covers diabetes and its complication, the role of diet, exercise, and medication, and the importance of self-monitoring. It is presented over 5 weeks where participants will learn and practice self-management skills, and help one another address family, cultural, or health system barriers to managing your diabetes. Following the 5-week curriculum, participants will be enrolled in the digital texting platform, Dulce Digital, in which they will receive on-going support via text messages derived from the curriculum, medication reminders, and blood glucose monitoring prompts in Tagalog.

SUMMARY:
This study aims to culturally adapt an existing American Diabetes Association (ADA)-recognized diabetes self-management and support or DSMES (Diabetes Self Management Education Support) program (Project Dulce) and integrate an evidence-based text messaging program (Dulce Digital) for implementation in Filipino Americans (FAs) with type 2 diabetes mellitus (T2DM). Cultural adaptations aims to facilitate and enhance patient centered approaches and increase participant engagement by addressing barriers to DSMES unique to FAs, such as linguistic challenges, health literacy and numeracy, cultural beliefs and values, and technology access and use. In addition, this study aims to examine the effectiveness of the culturally and digitally adapted Project Dulce + Dulce Digital in improving diabetes knowledge, belief, attitudes, hemoglobin A1C (glycosylated hemoglobin), and self-management behaviors at baseline to 3 months and 6 months. The unprecedented increase of T2DM prevalence among racial and ethnic minority populations including FAs in recent decades demands for effective strategies to meet the needs in DSMES in this population. The outcomes of the current study will demonstrate that the culturally adapted Project Dulce and integration of Dulce Digital is effective in addressing the needs FAs, an underserved racial and ethnic minority group in high need of culturally appropriate DSMES.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) disproportionately affects racial and ethnic minority populations. Among Asian Americans, Filipino Americans (FA) have the second highest T2DM prevalence and have an increased risk for developing complications due to lack of engagement in health protective behaviors (e.g., eating healthfully, obtaining adequate activity) and increased social and environmental barriers to optimal self-management (e.g., access to culturally appropriate education programs). While diabetes self-management education (DSME) programs have been shown to significantly improve T2DM outcomes, fewer than 10% of newly-diagnosed individuals receive DSMES within the first year of diagnosis.

Project Dulce is an American Diabetes Association (ADA)-recognized adult T2DM management program developed to address the needs of a racially and ethnically diverse San Diego population. Project Dulce includes a multi-disciplinary team with peer educators delivering DSMES. Previous trials have shown Project Dulce team-care improves clinical management and reduces costs (e.g., Philis-Tsimikas et al., 2004; Gilmer et al., 2005), and that the peer education alone improves clinical outcomes in Hispanics with T2DM (Philis-Tsimikas et al., 2011). The program has been disseminated locally, nationally, and internationally to White and Hispanic populations and has now served over 20,000 people. More recently, the peer education content was adapted via the Dulce Digital program to extend the reach of the care team through text messages derived from the Project Dulce curriculum, including medication reminders, and blood glucose monitoring prompts. This program led to a significant reduction of hemoglobin AHbA1c across 10 months versus usual care in Hispanics with diabetes (Fortmann et al., 2017). While Project Dulce has been adapted and demonstrated improvements in clinical and cost outcomes in Hispanic patients, cultural and digital adaptations are needed to increase and facilitate use in other racial and ethnic minority groups including FAs.

Using a Community-Based Participatory Research (CBPR) approach, this study will adapt Project Dulce + Dulce Digital for implementation in FA adults with T2DM. Cultural adaptations aims to facilitate and enhance patient-centered approaches by addressing barriers to DSMES unique to this population, such as linguistic challenges, health literacy and numeracy, cultural beliefs and values, and technology access and use. In addition, ADA has recommended the use of digital technologies as effective methods to deliver DSMES and mitigate barriers to participation. The adaptation process will be demonstrated in partnership with a local Federally Qualified Health Center (FQHC) serving a large number of FAs from diverse socioeconomic backgrounds. This study aims to culturally adapt Project Dulce and Dulce Digital for FAs with T2DM. Specifically, this study aims to:

1. examine the effectiveness of the culturally adapted Project Dulce + Dulce Digital in improving diabetes knowledge, attitudes, and beliefs among FAs with T2DM;
2. examine the effectiveness of the culturally adapted Project Dulce + Dulce Digital in improving HbA1C and self-management behaviors (i.e., diet, physical activity, medication adherence, foot care, blood glucose monitoring from baseline to 3- and 6-months; and
3. evaluate the acceptability and feasibility of the culturally adapted Project Dulce + Dulce Digital when delivered by FA peer educator to FA patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Filipino
* Diagnosed with T2DM
* Registered at Scripps Health or San Ysidro Health (or willing to register)
* HbA1c ≥7.5% and/or systolic blood pressure ≥ 140, and/or LDL-C ≥ 100 mg/dL within 90 days
* Able to speak, read, write, and comprehend in English and Tagalog
* Have access to a cell phone that can receive/send text messages throughout the study

Exclusion Criteria:

* Severe illness precluding frequent visits to clinic
* Liver function tests (ALT and AST) > 3 times the upper limit of normal
* Body mass index ≤ 23 kg/cm
* History of malignancy, except subjects who have been disease-free for >years, or whose only malignancy has been basal or squamous cell skin carcinoma
* Creatinine >3.5
* History of drug or alcohol abuse within 12 months prior to enrollment
* Not a permanent resident in the area
* Current enrollee in Project Dulce
* Blood donation of one pint or more within the past 30 days, or plasma donation within 7 days prior to screening
* Anemia
* Type 1 or gestational diabetes
* Pregnant
* Are currently participating in another diabetes-related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Diabetes Knowledge at 3 months | 3 months
  Diabetes Knowledge Test (Fitzgerald, Funnell, Anderson, et al., 2016) is a 23-item measure of diabetes knowledge, with general questions related to symptoms, self-management (e.g., diet, exercise, foot care, blood glucose monitoring, insulin) , and complications (e.g., low and high blood sugar). Greater scores indicate greater diabetes knowledge.
Change from Baseline Diabetes Knowledge at 6 months | 6 months
  Diabetes Knowledge Test (Fitzgerald, Funnell, Anderson, et al., 2016) is a 23-item measure of diabetes knowledge, with general questions related to symptoms, self-management (e.g., diet, exercise, foot care, blood glucose monitoring, insulin) , and complications (e.g., low and high blood sugar). Greater scores indicate greater diabetes knowledge.
Change in Baseline Self-Efficacy for Diabetes Scale at 3 months | 3 months
  Stanford Self-Efficacy for Diabetes Scale (Lorig, Stewart, Ritter, et al., 1996) is comprised of 8 items that measure the confidence of a participant in performing self-care activities such as eating meals every 4 to 5 hours, following a healthful diet, exercising, and blood glucose monitoring. Response options range from 1=not at all confident to 10=totally confident, with higher scores indicating greater self-efficacy.
Change in Baseline Self-Efficacy for Diabetes Scale at 6 months | 6 months
  Stanford Self-Efficacy for Diabetes Scale (Lorig, Stewart, Ritter, et al., 1996) is comprised of 8 items that measure the confidence of a participant in performing self-care activities such as eating meals every 4 to 5 hours, following a healthful diet, exercising, and blood glucose monitoring. Response options range from 1=not at all confident to 10=totally confident, with higher scores indicating greater self-efficacy.

SECONDARY OUTCOMES:
Change in Baseline Summary of Diabetes Self-Care Activities at 3 months | 3 months
  Summary of Diabetes Self-Care Activities measure (Toobert, Hampson, & Glassgow, 2000) is a 13-item brief questionnaire that assesses respondents adherence to self-management behavior recommendations in the past 7 days, including general and specific diet, exercise, blood glucose testing, foot care, medication adherence, and smoking, with greater scores indicating greater adherence.
Change in Baseline Summary of Diabetes Self-Care Activities at 6 months | 6 months
  Summary of Diabetes Self-Care Activities measure (Toobert, Hampson, & Glassgow, 2000) is a 13-item brief questionnaire that assesses respondents adherence to self-management behavior recommendations in the past 7 days, including general and specific diet, exercise, blood glucose testing, foot care, medication adherence, and smoking, with greater scores indicating greater adherence.
Change in Baseline Block Food Frequency Questionnaire at 3 months | 3 months
  Block Food Frequency Questionnaire (Block et al., 1995) measures frequency of fruit, vegetable and fiber consumption, and fat (and saturated fat) consumption each week using seven frequency categories ranging from less than once a week to 2 or more a day. Minor modifications were included to add food items commonly consumed in a Filipino diet (e.g., "Any other vegetables such as corn broccoli, zucchini, or vegetables commonly used Filipino cooking such as sitaw, kalabasa, sayote, upo, monggo, malunggay, amapalaya, pechay, kangkong, okra, etc.)
Change in Baseline Block Food Frequency Questionnaire at 6 months | 6 months
  Block Food Frequency Questionnaire (Block et al., 1995) measures frequency of fruit, vegetable and fiber consumption, and fat (and saturated fat) consumption each week using seven frequency categories ranging from less than once a week to 2 or more a day. Minor modifications were included to add food items commonly consumed in a Filipino diet (e.g., "Any other vegetables such as corn broccoli, zucchini, or vegetables commonly used Filipino cooking such as sitaw, kalabasa, sayote, upo, monggo, malunggay, amapalaya, pechay, kangkong, okra, etc.)
Change in Baseline International Physical Activity Questionnaire-Short Form at 3 months | 3 months
  International Physical Activity -Short Form (Craig et al., 2003) assesses the amount of physical activity (work, leisure, and other) and sedentary time in the past 7 days.
Change in Baseline International Physical Activity Questionnaire-Short Form at 6 months | 6 months
  International Physical Activity -Short Form (Craig et al., 2003) assesses the amount of physical activity (work, leisure, and other) and sedentary time in the past 7 days.
Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 3 months; % Units | 3 months
  HbA1c is measure of blood sugar level and assessed using blood samples following a 12-hour fast. Samples will be processed by Quest Diagnostics Inc and assayed by Immunoturbidimetry (Integra 800, Roche).
Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 6 months; % Units | 6 months
  HbA1c is measure of blood sugar level and assessed using blood samples following a 12-hour fast. Samples will be processed by Quest Diagnostics Inc and assayed by Immunoturbidimetry (Integra 800, Roche).

OTHER OUTCOMES:
Recruitment and Retention | 6 months
  Recruitment rate is the number of participants recruited divided by the maximum number of sites (n=1), divided by the number of months recruiting.
  Retention rate is the number of participants who remained in the study at the last wave of data collection (6 months) as the proportion of the number of participants enrolled at the baseline assessment.
Participant Satisfaction | 6 months
  Study-adapted focus group questionnaire evaluates participant experiences and satisfaction related to specific aspects of the peer-led diabetes education program (e.g., curriculum, handouts and PowerPoint Slides, peer educator) and text messaging component (e.g., content of text messages, receiving and responding to text messages, follow-up phone calls from the peer educator).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rose N. San Diego, PhD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (2):
- United States (2):
  - San Ysidro Health, National City, California
  - Scripps Whittier Diabetes Institute, San Diego, California

IPD SHARING:
Plan to Share IPD: No